CLINICAL TRIAL: NCT05505370
Title: Case Series With Saneso 3600 Colonoscope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saneso Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SAN360LGICL
Record Dates: First submitted 2022-08-16; First posted 2022-08-17 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Colonic Neoplasms
Keywords: Colonoscopy; Colonoscope
MeSH Terms: conditions — Colonic Neoplasms | interventions — Colonoscopy

STUDY DESIGN:
Intervention Model Description: The objective of the present study is to Study the clinical success and clinical safety of the Saneso colonoscope
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Study Arm Study device (Experimental): Patients who meet all eligibility criteria were included and had a clinically indicated colonoscopy procedure performed using the study device. Immediately thereafter, patients had a colonoscopy procedure using standard colonoscope (Olympus CF 180) by a second endoscopist.
  Interventions: Device: Colonoscopy
- Study Arm - Predicate Device (Active Comparator): Patients who meet all eligibility criteria were included and had a clinically indicated colonoscopy procedure performed using the study device. Immediately thereafter, patients had a colonoscopy procedure using standard colonoscope (Olympus CF 180) by a second endoscopist.
  Interventions: Device: Colonoscopy

INTERVENTIONS:
Device: Colonoscopy — Patients who meet all eligibility criteria were included and had a clinically indicated colonoscopy procedure performed using the study device. Immediately thereafter, patients had a colonoscopy procedure using standard colonoscope (Olympus CF 180) by a second endoscopist.

SUMMARY:
Saneso colonoscope is a novel FDA cleared colonoscope that provides a 360 degree integrated view of the colon. Saneso colonoscope has five cameras and multiple LED lights at the distal head. The objective of the present study is to evaluate clinical success of the Saneso colonoscope in intubation of the terminal ileum and to obtain user feedback with regards to usability characteristics compared to predicate devices.

DETAILED DESCRIPTION:
This study is a prospective, multi-center case series of per standard of care colonoscopy procedures using a nonsignificant risk Saneso 360 degree colonoscope. 40 cases were included at 3 clinical sites. Patients who meet all eligibility criteria were included and had a clinically indicated colonoscopy procedure performed using the study device. Immediately thereafter, patients had a colonoscopy procedure using standard colonoscope (Olympus CF 180) by a second endoscopist. Enrolled subjects were followed for 7 days after their procedure. If the procedure was not successful with the study device, the endoscopist completed the procedure with a traditional colonoscope used at each facility. This study was approved by the institutional review board of respective sites. The clinical trial was conducted in accordance with the standards of Good Clinical Practice (GCP) and in accordance with the principles of the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* 45 -74 years of age Willing and able to comply with the study procedures and provide written informed consent to participate in the study.

Scheduled for a clinically indicated routine colonoscopy procedure ASA class 1-3.

Exclusion Criteria:

* Altered colon anatomy Pregnant women, children under 18 years of age and adults over 75 years of age. Subjects for whom routine endoscopic procedures are contraindicated due to comorbid medical conditions.

Patients who are currently enrolled in another investigational study that would directly interfere with the current study, without prior written approval from the sponsor ASA class 4-5.

Ages: 45 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Intubation of terminal ileum and cecum | 4 months.
  Intubation of the terminal ileum and cecum

SECONDARY OUTCOMES:
User feedback for operating characteristics of the device | 4 months.
  User feedback for operating characteristics of the device

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Valley Endoscopy Center, Saint Clairsville, Ohio
  - Wintersville Endoscopy Center, Wintersville, Wintersville, Ohio
  - West Virginia University School of Medicine - Davis Medical Center, Elkins, West Virginia
  - West Virginia University School of Medicine - Reynolds Memorial Hospital, Glendale, West Virginia
  - West Virginia University School of Medicine - Reynolds Memorial Hospital,, Glendale, West Virginia